CLINICAL TRIAL: NCT01687504
Title: Pharmacokinetics and Safety of the WHO Recommended Increased Dosages of the First-line Anti-TB Medications in Children With TB and HIV/TB Coinfection
Brief Title: Pharmacokinetics of Anti-TB Drugs in HIV/TB Co-infected Children in Ghana
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PK-PTBHIV01; R01HD071779 (NIH)
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-09

CONDITIONS: Tuberculosis; HIV
Keywords: pharmacokinetics; children; HIV; Tuberculosis; Pharmacogenetics
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA plasma for analysis of drug concentrations Whole blood DNA for for genotyping of drug metabolizing enzymes and transporters
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Tuberculosis (also known as TB) is a common infection and a major cause of death in children. Effective treatment using a combination of anti-tuberculosis (anti-TB) medications saves lives, but dosages of these medications are not well established in children. Several research studies have shown that the recommended dosages of the anti-TB medications in children do not lead to adequate blood levels to kill the bacteria in some children. This situation may lead to treatment failure and emergence of drug resistance. As a result, the world Health Organization (WHO) recently recommended increased dosages for all the TB medications in children. This study is being conducted to find out if the increased dosages of the anti-TB drugs are safe and lead to adequate drug levels in the blood of children with TB with or without HIV infection.

DETAILED DESCRIPTION:
The treatment guidelines for childhood TB are largely inferred from studies in adults, as few controlled trials have been done in children to establish optimum regimens. The standard anti-TB treatment consists of a combination of isoniazid, rifampin, pyrazinamide and ethambutol for two months induction phase followed by 2 months of isoniazid and rifampin in the continuation phase. The plasma and tissue concentrations of each of the drugs in the combination regimen needs to be optimized to maximize bacterial killing and reduce the risk of treatment failure with emergence of drug resistance. Several studies have shown that the peak concentrations of these drugs in a large proportion of children are so low that there is a concern for ineffective therapy in some children. This concern led to the recent recommendation by the WHO to increase the dosages of all first-line anti-TB drugs in children. To our knowledge, the safety and pharmacokinetics of the new dosages have not been studied in children in West Africa. In addition, differences in drug absorption, metabolism and excretion may put some children at risk of low drug concentrations when the standard weight-based fixed-dosages are prescribed to all children. Identification of these individuals clinically or through genetic testing may be important for individualized dosing. The factors that may influence drug concentrations and treatment effects include age, HIV coinfection status, nutritional status and genetic polymorphisms of drug metabolizing enzymes and transporters. Younger children appear to eliminate the drugs faster and have lower plasma peak concentrations compared to older children and adults treated with similar mg/kg doses. The association between nutritional status and the plasma pharmacokinetics of the anti-TB drugs is less clear, as some but not all studies report a significant relationship. HIV coinfection is an important factor that has been associated with poor treatment responses as a result of poor drug absorption.

The primary objective of this study is to evaluate the pharmacokinetics and tolerability of the elevated dosages of the first-line anti-TB in children, as well as factors associated with inter-individual variability in anti-TB drugs exposure in Ghanaian children.

A two-arm pharmacokinetic study in children with active TB with or without HIV coinfection will be performed at Komfo Anokye Teaching Hospital, Kumasi, Ghana. Children aged between 3 months and 14 years, for whom informed consent by parent or guardian have been obtained, will be enrolled. A complete medical history, physical examination, and nutritional status assessment will be performed at enrolment at subsequent study visits. Relevant data will be collected using standardized forms. Baseline measurements prior to initiation of anti-TB treatment will include complete blood count (CBC), blood urea nitrogen, creatinine, liver function tests (LFTs), as well as CD4 cell count determination and plasma HIV-1 RNA level (if HIV co-infected). Measurements LFTs will be repeated at week 2 of therapy or when clinically indicated to evaluate for drug toxicity. All study participants will follow-up at 2 and 4 weeks and then monthly to assess adverse events and clinical response to therapy.

Anti-TB treatment will be initiated immediately upon TB diagnosis and concurrent initiation ART will be allowed in co-infected children as per national and WHO guidelines. The standard anti-TB regimen consists of daily ingestion of isoniazid, rifampin, pyrazinamide and ethambutol for 2 months, then rifampin and isoniazid daily for 4 months. The new WHO recommended doses for children will be prescribed. Weight-based fixed-dose combination tablets are used. Children will receive directly observed therapy for the anti-TB treatment by healthcare worker at the hospital or family member at home. Treatment outcome (completed/cured, died, defaulted, discontinued, transferred out) is defined according to WHO criteria.

Pharmacokinetic sampling will be performed at 4 weeks of anti-TB therapy. Study drugs will be administered after at least a 2-hour fast in non-breastfed children and blood samples obtained through intravascular catheters at times 0, 2, 4, 6, 8-hours post dosing. Actual times of dosing and sampling will be accurately recorded. Doses vomited < 30 minutes after dosing will require cancellation of PK testing and rescheduling. The samples will be placed immediately on ice and centrifuged within 30 minutes at 3000g for 10 minutes at 4oC. Plasma will be stored at - 70oC until measurement of drug concentrations. Drug concentrations will be determined using validated gas chromatography with mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

1. Children with active TB with or without HIV co-infection. Active TB diagnosis defined by clinical criteria consistent with active TB and/or a positive AFB smear or mycobacterial culture.
2. Aged 3 months to 14 years old.
3. Available for follow-up until completion of TB treatment and/or achievement of a study endpoint like discontinuation of therapy, and/or pharmacokinetic sampling.

Exclusion Criteria:

1. Unable to obtain informed signed consent parent(s) or legal guardian.
2. Have AIDS-related opportunistic infections other than TB, history of or proven acute hepatitis within 30 days of study entry, persistent vomiting, or diarrhea.
3. Hemoglobin < 6 g/dl, white blood cells < 2500/mm3, serum creatinine > 1.5 mg/dl, AST and ALT > 2X upper limit of normal.

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3 months to 14 years old with active tuberculosis with or with HIV coinfection
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Descriptive statistics of PK parameters (Cmax, Tmax, AUC0-8h) of rifampin, isoniazid, pyrazinamide and ethambutol in children with TB with and without HIV coinfection | Week 4 of therapy

SECONDARY OUTCOMES:
Frequency of liver enzymes elevations compare to baseline, skin rashes, nausea, vomiting and treatment discontinuation or modifications due to drug side effects in children with TB with and without HIV coinfection | up to week 24
  The frequency of each drug side effects between children with TB and children with with HIV/TB confection on standard anti-TB therapy will be compared by chi-square test
Relationship between genetic polymorphisms of N-acetyltransferase type 2 (NAT2) enzyme and isoniazid plasma Cmax and AUC in Ghanaian children with TB with and without HIV | Week 4 of therapy
  Genetic effect of each genetic variant on PK parameter will be estimated as odds ratio between carrier and non-carrier for each variant
Relationship between genetic polymorphisms of SLCO1B1 transporter and rifampin plasma Cmax and AUC in Ghanaian children with TB with and without HIV | week 4 of therapy
  Genetic effect of each genetic variant on PK parameter will be estimated as odds ratio between carrier and non-carrier for each genetic variant
Relationship between plasma Cmax and AUC of isoniazid, rifampin, ethambutol and pyrazinamide at week 4 of therapy and frequency of anti-TB treatment discontinuation or modification | up to week 24
  Differences in mean Cmax and AUC of each drug between children who complete 6 months anti-TB therapy and those who require treatment modification due to drug side effects will be compared by t-test or non-parametric test. Note that treatment modification due to drug side effects is as per national TB treatment guidelines but no new interventions are prescribed in this observation study.
Relationship between NAT2 acelator status, SLCO1B1 genotype status and anti-TB treatment completion, discontinuation or modification | up to week 24
  Genetic effect of each genetic variant on treatment discontinuation or modification rates will be estimated as odds ratio between carrier and non-carrier for each variant. Note that treatment modification due to drug side effects is as per national TB treatment guidelines but no new interventions are prescribed in this observation study.
Relationship between body weight, gender, nutritional status and plasma Cmax and AUC of isoniazid, rifampin, ethambutol and pyrazinamide in Ghanaian children with TB with and without HIV | up to week 4 of therapy
  Appropriate regression model will be used to test correlation between clinical factors and anti-TB drugs PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Awewura Kwara, MD, MPH&TM, Principal Investigator — The Miriam Hospital
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ghana

REFERENCES:
- [Derived] Horita Y, Alsultan A, Kwara A, Antwi S, Enimil A, Ortsin A, Dompreh A, Yang H, Wiesner L, Peloquin CA. Evaluation of the Adequacy of WHO Revised Dosages of the First-Line Antituberculosis Drugs in Children with Tuberculosis Using Population Pharmacokinetic Modeling and Simulations. Antimicrob Agents Chemother. 2018 Aug 27;62(9):e00008-18. doi: 10.1128/AAC.00008-18. Print 2018 Sep. PMID 29914960
- [Derived] Antwi S, Yang H, Enimil A, Sarfo AM, Gillani FS, Ansong D, Dompreh A, Orstin A, Opoku T, Bosomtwe D, Wiesner L, Norman J, Peloquin CA, Kwara A. Pharmacokinetics of the First-Line Antituberculosis Drugs in Ghanaian Children with Tuberculosis with or without HIV Coinfection. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e01701-16. doi: 10.1128/AAC.01701-16. Print 2017 Feb. PMID 27855070